CLINICAL TRIAL: NCT01921829
Title: Effect of Protocolized Diuretic Strategy on Clinical Outcomes and Health-related Quality of Life in Cardiorenal Failure: A Randomized Trial
Brief Title: Protocolized Diuretic Strategy in Cardiorenal Failure
Acronym: ProDiuS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to futility due to lower than expected recruitment
Sponsor: Kelly V. Liang, MD (Other)
Responsible Party: Sponsor-Investigator, Kelly V. Liang, MD, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO13040071
Record Dates: First submitted 2013-07-23; First posted 2013-08-13 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Cardiac Failure; Renal Failure; Kidney Failure
Keywords: Cardiorenal failure; Cardiorenal syndrome; Diuretic resistance; Volume overload; Edema; Health-related quality of life; Outcomes; Treatment protocol
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardio-Renal Syndrome; Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Participants randomized to the Usual Care group (control arm) will receive escalating diuretics and medical therapy per HF guidelines published by the American College of Cardiology (ACC)/American Heart Association (AHA) and Heart Failure Society of America (HFSA), dosed in variable fashion at the discretion of the treating cardiologist.
- Protocolized Diuretic Strategy (Experimental): Participants randomized to the Protocolized Diuretic Strategy group will receive escalating diuretics according to an algorithm targeting a goal diuresis of urine output (UO) 3-5 L/day with diuretics intensified in a stepped fashion using both loop diuretics given by intravenous (IV) bolus followed by IV continuous infusion (furosemide or alternative loop diuretic at equivalent dose), with or without concomitant thiazide diuretic (oral (PO) metolazone or IV chlorothiazide). If UO is < 3 L/day, diuretic regimen will be increased. If UO is 3-5 L/day, diuretic regimen will be continued at current doses. If UO is > 5 L/day, diuretic regimen will be reduced.
  Interventions: Drug: Protocolized Diuretic Strategy

INTERVENTIONS:
Drug: Protocolized Diuretic Strategy — The Protocolized Diuretic Strategy will administer diuretics according to an algorithm based on based on the "stepped pharmacologic care arm" used by the CARRESS-HF trial investigators. This algorithm targets a relatively aggressive goal diuresis of urine output (UO) 3-5 L/day with diuretics intensified in a stepped fashion using both loop diuretics given by intravenous (IV) bolus followed by IV continuous infusion (furosemide or alternative loop diuretic at equivalent dose), with or without concomitant thiazide diuretic (oral (PO) metolazone or IV chlorothiazide).
  Other Names: Diuretic Treatment Protocol; Stepped Pharmacologic Care
  Arms: Protocolized Diuretic Strategy

SUMMARY:
This research study is a randomized clinical trial to evaluate if taking diuretics (medications that increase urine production and help with fluid removal from the body) in a standardized fashion (using a guideline for adjusting doses based on measured urine output) could improve health outcomes in patients with cardiorenal failure or cardiorenal syndrome (combined heart and kidney failure) with edema (too much fluid in their arms, legs, and/or lungs). Under usual care, these patients are treated with diuretics and other medications in increasing doses, but not necessarily to maintain a specific amount of urine output per day. Current heart failure (HF) treatment guidelines do not provide any standard protocol, or guideline, for adjusting diuretic doses. At the point when kidney function worsens to the degree that the kidneys are no longer able to respond to the medications used to remove fluid, either ultrafiltration (UF) or dialysis (also called hemodialysis [HD]) is typically started in order to remove fluid. In both UF and dialysis, excess fluid is removed from the body by using a machine. In dialysis, both waste products and fluid are removed and electrolyte abnormalities are corrected. In UF, only fluid is removed. Both procedures use the same machine. This study will test whether a Protocolized Diuretic Strategy (ProDiuS), a plan for adjusting diuretic doses based on measured urine output, will improve clinical care for cardiorenal syndrome. Such a plan for adjusting diuretic doses is needed to improve symptoms, decrease the length of hospital stays and rehospitalization rates, and improve health-related quality of life (HRQOL) in cardiorenal syndrome patients.

DETAILED DESCRIPTION:
Heart failure (HF) accounts for over 1 million hospital admissions annually in the United States and is a leading cause of disability and healthcare costs. Cardiorenal syndrome and worsening renal function are independent risk factors for morbidity and mortality in HF. Effective fluid removal, manifested by a decrease in body weight, is one of the most important goals of treatment in cardiorenal syndrome. Current medical therapeutic options, including sodium and fluid restriction, diuretics, blockade of the renin-angiotensin-aldosterone system, inotropes, and nesiritide, are suboptimal in patients with advanced cardiorenal syndrome. When medical therapies fail, ultrafiltration (UF) may be used for mechanical fluid removal using dialysis or UF machines. UF can effectively remove fluid in HF patients, but its precise role in the therapy of cardiorenal syndrome is still unclear. A multicenter randomized controlled trial (CARRESS-HF) suggested that UF was not superior to a stepped pharmacologic diuretic regimen, with a similar amount of weight loss with the two approaches and a higher rate of adverse events in the UF group. Therefore, a protocolized diuretic strategy is needed that is superior to current clinical care in the management of cardiorenal syndrome.

Current HF guidelines do not provide any standard protocol for diuretic dosing. The variation in usual clinical care may explain the long hospital stays and worsening renal function common in these patients. One retrospective observational study compared a diuretic dosing protocol to usual diuretic therapy for patients admitted with acute decompensated HF. Protocol diuretic use was associated with greater weight loss and significantly lower risk of 30-day readmission. However, due to its retrospective design, the baseline characteristics of the two groups differed in many pertinent covariates, and its generalizability is limited.

The proposed study aims to determine if a protocolized diuretic treatment strategy, as opposed to usual clinical care, results in improved clinical decongestion, clinical outcomes, and health-related quality of life (HRQOL), while preserving renal function in hospitalized patients with cardiorenal syndrome. It is a prospective randomized single-blind trial with equal allocation (1:1) and random block randomization of 150 participants hospitalized at University of Pittsburgh Medical Center (UPMC) for cardiorenal syndrome recruited over 3 years (approximately 50 participants/year). Participants with cardiorenal syndrome will be randomized to a Protocolized Diuretic Strategy (based on the stepped pharmacologic algorithm used in the CARRESS-HF trial) vs. Usual Care. Participants will be followed daily in the hospital during the treatment period, as well as at 1-month and 3-month follow-up visits in the outpatient HF clinic.

Primary Research Question:

1. In hospitalized patients with cardiorenal syndrome, does a protocolized diuretic treatment strategy, as opposed to usual clinical care, result in improved clinical decongestion based on change in body weight at day 4 or hospital discharge (whichever comes first)? Primary Hypothesis. In hospitalized patients with cardiorenal syndrome, protocolized diuretic therapy will result in greater reduction in body weight and improved clinical decongestion compared to usual care.

Secondary Research Questions:

1. Do clinical outcomes, including length of hospitalization, number of rehospitalizations for HF, and mortality, improve after protocolized diuretic therapy compared to usual care over 3 months? Hypothesis 1. Protocolized diuretic therapy will be associated with reduced length of hospital stay, decreased rehospitalization rates, and decreased mortality, compared to usual care.
2. Do other measures of volume status improve after protocolized diuretic therapy compared to usual care during hospitalization and over 3 months? Hypothesis 2. Protocolized diuretic therapy will be associated with greater decongestion based on increased venous compliance of the internal jugular vein (via Doppler ultrasound), negative fluid balance, and clinical decongestion, compared to usual care.
3. Do HRQOL outcomes improve after protocolized diuretic therapy compared to usual care over 3 months? Hypothesis 3. HRQOL indices in physical well-being, mental well-being, and sleep quality domains will improve after protocolized diuretic therapy compared to usual care.
4. Do renal outcomes (safety endpoints), including renal function changes and need for UF or renal replacement therapy, differ between protocolized diuretic therapy and usual care during hospitalization and over 3 months? Hypothesis 4. Protocolized diuretic therapy will be superior to usual care in terms of worsening renal function and need for UF or renal replacement therapy.

Subgroup Research Questions:

1. Do outcomes differ between the Protocolized Diuretic Strategy vs. Usual care stratified by type of heart failure (e.g., systolic dysfunction (EF <40%) vs. diastolic dysfunction (EF ≥40%); ischemic vs. other; none-mild vs. moderate-severe mitral regurgitation (MR) or tricuspid regurgitation (TR))? Hypothesis 1. No difference will be seen between treatment and control groups based on type of heart failure.

This trial is of utmost interest to cardiologists and nephrologists, who struggle to find the optimal diuretic and medical management strategy to effectively remove excess fluid yet preserve renal function. It is highly relevant to many clinicians and the community at large, as HF and cardiorenal syndrome are a leading cause of hospitalizations and healthcare costs. If a protocolized diuretic strategy can be found that optimally removes fluid in an efficient and safe manner, it could potentially be disseminated to community physicians and/or incorporated into public policy or HF treatment guidelines in order to improve quality of care and reduce healthcare costs in this population with high morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* History of heart failure (HF), with either left ventricular (LV) dysfunction (EF<40%) or at least stage I diastolic or right ventricular (RV) dysfunction based on echocardiogram (ECHO) within the last year or diagnosis of HF by International Classification of Diseases (ICD-9)
* Evidence of renal dysfunction based on one of the following:

  * Estimated glomerular filtration rate (GFR) 15-59 mL/min/1.73 m2 based on the Modification of Diet in Renal Disease (MDRD) equation using serum creatinine (Cr) obtained within 6 months of admission
  * Elevated Cr above upper limits of normal
  * An increase in serum Cr of ≥0.3 mg/dL or ≥50% from baseline on admission or during diuretic therapy, with no alternative cause for worsening renal function, while demonstrating signs and symptoms of persistent volume overload occurring within 7 days before admission or during hospitalization
* Evidence of volume overload by clinical and/or radiographic features, with at least 2 of the following: 1) peripheral edema ≥2+; 2) jugular venous distension ≥7 cm; 3) radiographic pulmonary edema or pleural effusion; 4) enlarged liver or ascites; 5) pulmonary rales, paroxysmal nocturnal dyspnea, or orthopnea; 6) elevated brain natriuretic peptide (BNP) level; 7) documentation of elevated right heart filling pressures by pulmonary artery catheter or right heart catheterization

Exclusion Criteria:

* Use of inotropes (at time of screening)
* Acute indications for hemodialysis (HD) (e.g., severe hyperkalemia, metabolic acidosis, uremic signs or symptoms, pericardial friction rub)
* Specific forms of HF by chart diagnoses:

  1. Congenital heart disease
  2. Primary valvular heart disease due to severe valvular stenosis or acute severe valvular regurgitation or valvular disease requiring immediate surgical repair
  3. Infiltrative cardiomyopathies
  4. Pulmonary hypertension (PH) as defined by World Health Organization (WHO) group I and WHO group IV - Prior use of ultrafiltration (UF) or HD in the 3 months preceding hospitalization
* End-stage renal disease (ESRD) requiring chronic dialysis or estimated GFR <15 mL/min/1.73 m2 by MDRD equation (i.e., pre-existing ESRD)
* Prior cardiac or kidney transplantation
* Intravascular volume depletion based on clinical assessment
* Cardiogenic shock and/or systolic blood pressure (SBP) <90 mmHg
* Unstable coronary disease or acute coronary syndrome within 1 month of admission
* Alternative explanation for worsening renal function (e.g., obstructive nephropathy, contrast-induced nephropathy, acute tubular necrosis, intrinsic renal diseases)
* Life expectancy < 3 months due to other chronic health conditions (e.g., end-stage liver disease, pulmonary disease, malignancy, etc.)
* Psychiatric disorder requiring admission to a psychiatric hospital during HF admission
* Previous enrollment in this trial or other diuretic or UF trial in the prior 3 months
* Expected geographic unavailability for 3 months following hospital admission
* Pregnancy
* Inability to provide informed consent
* Physician's assessment that use of the protocol could be unsafe or lead to adverse consequences for the patient

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly V Liang, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Bart BA, Goldsmith SR, Lee KL, Givertz MM, O'Connor CM, Bull DA, Redfield MM, Deswal A, Rouleau JL, LeWinter MM, Ofili EO, Stevenson LW, Semigran MJ, Felker GM, Chen HH, Hernandez AF, Anstrom KJ, McNulty SE, Velazquez EJ, Ibarra JC, Mascette AM, Braunwald E; Heart Failure Clinical Research Network. Ultrafiltration in decompensated heart failure with cardiorenal syndrome. N Engl J Med. 2012 Dec 13;367(24):2296-304. doi: 10.1056/NEJMoa1210357. Epub 2012 Nov 6. PMID 23131078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the UPMC Heart Failure and Cardiology services, from July 2015-Nov 2016.
Pre-assignment Details: One participant was enrolled but withdrew consent before receiving any randomized treatment protocol. Therefore, that patient was withdrawn.
Period: Overall Study
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Protocolized Diuretic Strategy | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (8.6) | 68.4 (6.9) | 68.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Years of education [Mean (Standard Deviation); unit: years] | 13.5 (2.3) | 12.9 (2.4) | 13.2 (2.3)
Smoking [Count of Participants; unit: Participants]
  Current | 0 | 0 | 0
  Past | 5 | 6 | 11
  Never | 5 | 2 | 7
Alcohol use [Count of Participants; unit: Participants] | 1 | 2 | 3
Caffeine use [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 8 | 6 | 14
Cardiomyopathy type [Count of Participants; unit: Participants]
  Ischemic | 5 | 5 | 10
  Dilated | 1 | 2 | 3
  Hypertensive | 0 | 1 | 1
  Other | 4 | 0 | 4
NYHA Class [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Functional Classes:
  I - No limitation of physical activity. Ordinary physical activity does not cause heart failure (HF) symptoms like undue fatigue, palpitation, dyspnea (shortness of breath).
  II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in HF symptoms.
  III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity results in HF symptoms.
  IV - Unable to carry on any physical activity without discomfort. HF symptoms occur at rest and increase with any physical activity. Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 6 | 15
    II | 2 | 2 | 4
    III | 5 | 4 | 9
    IV | 2 | 0 | 2
Left ventricular ejection fraction [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 8 | 7 | 15
    20-25% | 3 | 2 | 5
    25-30% | 0 | 2 | 2
    30-35% | 1 | 0 | 1
    Unknown | 4 | 3 | 7
Right ventricular function [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 8 | 6 | 14
    Normal | 3 | 5 | 8
    Reduced | 5 | 1 | 6
Mitral regurgitation [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 7 | 6 | 13
    (all) | 4 | 3 | 7
Tricuspid regurgitation [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 8 | 6 | 14
    (all) | 6 | 4 | 10
Jugular venous pressure elevated [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 6 | 7 | 13
Edema grade [Count of Participants; unit: Participants] — Edema grades based on palpation of skin:
  1. - There is a barely detectable 2mm depression. Not easily seen but can be felt. Immediate rebound.
  2. - There is a 4mm deep pit. A few seconds to rebound.
  3. - There is a 6mm deep pit. 10-12 seconds to rebound.
  4. - There is an 8mm deep pit (very deep). >20 seconds to rebound. Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 7 | 16
    2+ | 7 | 2 | 9
    3+ | 1 | 3 | 4
    Unknown | 1 | 2 | 3
Hypertension [Count of Participants; unit: Participants] | 9 | 7 | 16
Diabetes mellitus [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 5 | 5 | 10
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 2 | 3 | 5
Coronary artery disease [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 5 | 6 | 11
Depression [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 2 | 2 | 4
Stroke [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 4 | 0 | 4
Peripheral vascular disease [Count of Participants; unit: Participants] | 4 | 0 | 4
Hyperlipidemia [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 5 | 5 | 10
Atrial fibrillation [Count of Participants; unit: Participants] | 5 | 6 | 11
Coronary artery bypass surgery [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 3 | 3 | 6
Implantable cardioverter defibrillator [Count of Participants; unit: Participants] | 5 | 2 | 7
Cardiac resynchronization therapy [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 1 | 1 | 2
Diuretic dose [Mean (Standard Deviation); unit: mg/day] — (furosemide equivalent)
  mg/day | 242.5 (112.7) | 166.3 (55.5) | 214.2 (99.7)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.9 (0.5) | 2.2 (0.8) | 2.0 (0.6)
Blood urea nitrogen [Mean (Standard Deviation); unit: mg/dL] | 38.2 (12.5) | 56.3 (38.8) | 45.6 (27.1)
Brain natriuretic peptide [Mean (Standard Deviation); unit: pg/mL] | 855.3 (690.7) | 530.4 (363.7) | 710.9 (578.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (kg) From Randomization to Day 4 or Date of Discharge (Whichever Comes First)
Description: The change in body weight (kg) from randomization to day 4 or date of discharge will be determined by the difference between body weight at day 4 after randomization or date of discharge (whichever comes first) and body weight taken at baseline measured in the hospital on standard scales without shoes and wearing a hospital gown, measured before breakfast and post-voiding.
Time Frame: 4 days (96 hours)
Population: One patient from ProDiuS arm withdrew before undergoing any randomized treatment.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
kg | -2.07 (4.84) | -6.12 (1.95)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.05, t-test, 2 sided

2. Secondary Outcome: Length of Hospitalization
Description: Length of hospitalization will be ascertained from admission date to date of discharge.
Time Frame: 1 month
Population: One participant from the ProDiuS arm withdrew consent before undergoing any randomized treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
days | 7.5 (12.0) | 8.0 (6.5)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.29, t-test, 2 sided

3. Secondary Outcome: Number of Rehospitalizations for Heart Failure (HF)
Description: Number of rehospitalizations for HF will be ascertained based on chart review of admissions with HF as a coded diagnosis, evidence of clinical volume overload, and treatment with intravenous diuretics.
Time Frame: Up to 3 months (assessed at 1 month and 3 months)
Measure: Number; unit: hospitalizations
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
hospitalizations | 3 | 1

4. Secondary Outcome: Number of Total Rehospitalizations
Description: Number of rehospitalizations will be ascertained based on chart review of admissions to any hospital after the index hospitalization
Time Frame: Up to 3 months (assessed at 1 month and 3 months)
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
hospitalizations | 0.0 (1.0) | 0.5 (5.5)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p > 0.95, Fisher Exact

5. Secondary Outcome: All-cause Mortality
Description: All-cause mortality will be ascertained based on chart review of vital status (alive/dead) and cause of death.
Time Frame: Up to 3 months (assessed at 1 month and 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 9
Participants | 1 | 4
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.58, Fisher Exact

6. Secondary Outcome: Difference From Baseline to 1 Month in Change in Right Internal Jugular Vein (RIJV) Cross-sectional Area (CSA) Pre- and Post-Valsalva
Description: The change in cross-sectional area (CSA) of the right internal jugular vein (RIJV) pre- and post-Valsalva is a measurement of venous compliance and was determined noninvasively with Doppler ultrasound. An increase in RIJV CSA >17% during Valsalva effectively rules out elevated right atrial pressure (RAP) and suggests effective volume removal or decongestion. The difference between baseline and 1 month values of change in RIJV CSA are reported.
Time Frame: Up to 1 month (measured at baseline and 1 mo)
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
cm^2 | 0.11 (1.03) | 0.22 (0.57)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.86, t-test, 2 sided

7. Secondary Outcome: Fluid Balance
Description: Strict intake (oral intake, intravenous medications, fluids, etc.) and output (urine, emesis, stools, drains, etc.) will be documented by the nurses on the HF floors per routine clinical protocol for all patients. Fluid balance will be determined by subtracting the volume of total intake from the volume of total output (in mL) over 24 hours (7 am to 7 am or the preceding 24-h period if no 7 am to 7 am period is available). Fluid balance and urine output will be ascertained by chart review daily during the intervention while the participants are hospitalized.
Time Frame: Daily while in hospital
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
mL/day | -1077 (345) | -590 (1268)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.40, t-test, 2 sided

8. Secondary Outcome: Acute Kidney Injury
Description: Acute kidney injury will be defined based a rise in Cr ≥0.3 mg/dL.
Time Frame: Daily while in hospital, 1 mo & 3 mos
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
Participants | 5 | 4
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p > 0.95, Fisher Exact

9. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Score Change at 1 Month
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a well-validated 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. A mean difference over time of 5 points on the KCCQ Overall Summary Scale reflects a clinically significant change in heart failure status. A 10 point decline in KCCQ scores has important prognostic significance in terms of survival.
Time Frame: Baseline to 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | 6.64 (18.01) | 19.89 (9.83)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.08, t-test, 2 sided

10. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Score Change at 1 Month
Description: as for outcome 9
Time Frame: Baseline to 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | 15.65 (14.41) | 16.20 (13.93)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p > 0.95, t-test, 2 sided

11. Secondary Outcome: SF-36 Mental Component Score (MCS) Change at 1 Month
Description: The Medical Outcomes Study (MOS) 36-item Short-Form Health Survey (SF-36) is a well-validated generic HRQOL questionnaire that generates two composite scores: the Physical Component Score (PCS) and Mental Component Score (MCS). The PCS aggregates items from Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, and Social Functioning. The MCS aggregates items from Role-Emotional, Mental Health, General Health, Vitality, and Social Functioning. The mean for each summary scale is 50 points with standard deviation of 10 points. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline to 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | -1.84 (15.41) | 4.96 (1.80)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.52, t-test, 2 sided

12. Secondary Outcome: SF-36 Physical Component Score (PCS) Change at 1 Month
Description: as for outcome 11
Time Frame: Baseline to 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | 12.31 (11.72) | 11.95 (11.40)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p > 0.95, t-test, 2 sided

13. Secondary Outcome: PHQ-9 Depression Index Change at 1 Month
Description: The Patient Health Questionnaire (PHQ-9) Depression Index is a well-established index of depression and has been validated in many patient populations. Its scores range from 0-27 with increasing scores representing increasing depression severity. Score categories represent depression severity and management recommendations:
  0-4 - Minimal or no depression. Monitor; may not require treatment. 5-9 - Mild. Use clinical judgment (symptom duration, functional impairment) to determine necessity of treatment.
  10-14 - Moderate. Use clinical judgment (symptom duration, functional impairment) to determine necessity of treatment.
  15-19 - Moderately severe. Warrants active treatment with psychotherapy, medications, or combination.
  20-27 - Severe. Warrants active treatment with psychotherapy, medications, or combination.
Time Frame: Baseline to 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | -3.5 (6.0) | -7.0 (10.0)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p > 0.95, t-test, 2 sided

14. Secondary Outcome: PSQI Total Score Change at 1 Month
Description: The Pittsburgh Sleep Quality Index (PSQI) is the most widely used global sleep assessment and has been studied in the renal transplant population. Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Traditionally, the items from the PSQI have been summed to create a total score to measure overall sleep quality.
Time Frame: Baseline to 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | -2.5 (5.0) | -1.0 (5.0)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.52, t-test, 2 sided

15. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Score Change at 3 Months
Description: as for outcome 9
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | 13.84 (17.04) | 24.47 (12.29)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.17, t-test, 2 sided

16. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Score Change at 3 Months
Description: as for outcome 9
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | 9.00 (17.24) | 23.00 (22.10)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.17, t-test, 2 sided

17. Secondary Outcome: SF-36 Mental Component Score (MCS) Change at 3 Months
Description: as for outcome 11
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | 6.06 (10.83) | -0.40 (0.62)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.40, t-test, 2 sided

18. Secondary Outcome: SF-36 Physical Component Score (PCS) Change at 3 Months
Description: as for outcome 11
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | 16.25 (8.50) | 12.90 (10.61)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p > 0.95, t-test, 2 sided

19. Secondary Outcome: PHQ-9 Depression Index Change at 3 Months
Description: The Patient Health Questionnaire (PHQ-9) Depression Index is a well-established index of depression and has been validated in many patient populations. Its scoring ranges from 0-27 with increasing scores representing increasing depression severity. Score categories determine depression severity and recommended management:
  0-4 - Minimal or none. Monitor; may not require treatment. 5-9 - Mild. Use clinical judgment (symptom duration, functional impairment) to determine necessity of treatment.
  10-14 - Moderate. Use clinical judgment (symptom duration, functional impairment) to determine necessity of treatment.
  15-19 - Moderately severe. Warrants active treatment with psychotherapy, medications, or combination.
  20-27 - Severe. Warrants active treatment with psychotherapy, medications, or combination.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | -1.00 (5.00) | -4.00 (7.50)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p = 0.55, t-test, 2 sided

20. Secondary Outcome: PSQI Total Score Change at 3 Months
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Traditionally, the items from the PSQI have been summed to create a total score to measure overall sleep quality.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
units on a scale | -1.00 (5.00) | -4.00 (8.00)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p > 0.95, t-test, 2 sided

21. Other Pre Specified Outcome: Adverse Events
Description: Hypokalemia (K <3.0 milliequivalents (mEq)/L), hypotension (systolic BP <90 mmHg), hyponatremia (Na <130 mEq/L), arrhythmias, cramps, and other (recorded as short description).
Time Frame: Daily while in hospital , 1 mo, & 3 mos
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Usual Care | Protocolized Diuretic Strategy
Number analyzed (Participants) | 10 | 8
events | 2.0 (6.0) | 3.5 (7.0)
Statistical Analysis 1: Comparison: Usual Care vs Protocolized Diuretic Strategy; Test type: Superiority; p > 0.95, Fisher Exact

ADVERSE EVENTS:
Time Frame: 3 months
Description: Acute kidney injury, hypokalemia (K <3.0 mEq/L), hypotension (systolic BP <90 mmHg), hyponatremia (Na <130 mEq/L), arrhythmias, cramps, and other were recorded. For each adverse event, diagnosis, date of onset, date of resolution, severity, whether it was unexpected, related to the intervention, serious adverse event (SAE), type of SAE, whether the blind was broken, and the outcome were recorded.
Arm/Group | Usual Care | Protocolized Diuretic Strategy
All-Cause Mortality (participants affected / at risk) | 1/10 | 4/9
Serious Adverse Events (participants affected / at risk) | 2/10 | 1/9
Other Adverse Events (participants affected / at risk) | 7/10 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=10) | Protocolized Diuretic Strategy (N=9)
Cardiac arrhythmia (Cardiac disorders) | 2 (4) | 1 (2)
Hospitalization (Cardiac disorders) | 2 (3) | 0 (0) — Volume overload or heart transplant
Hospitalization for non-cardiac cause (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Acute gout flare, leukocytosis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=10) | Protocolized Diuretic Strategy (N=9)
Hypokalemia (Renal and urinary disorders) | 3 (4) | 1 (1)
Hyponatremia (Renal and urinary disorders) | 4 (5) | 2 (2)
Hyperphosphatemia (Renal and urinary disorders) | 2 (2) | 0 (0)
Worsening acute kidney injury (Renal and urinary disorders) | 6 (9) | 1 (2)
Hypercalcemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypermagnesemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Hyperkalemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (2) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 0 (0) | 1 (1) — Hitting head on wall
Severe head/neck pain (General disorders) | 1 (1) | 0 (0)
Leg and abdominal cramps (General disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — High depression score requiring follow up from psychiatry

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No